CLINICAL TRIAL: NCT03232190
Title: The Use of an Age-linked Web Application for Parents During and After a NICU Stay in Improving Child Development and Parent Empowerment
Brief Title: The Use of an Age-linked App for Parents During and After a NICU Stay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: KU Leuven (Other); TRACE: Centre For Translational Psychological Research (Unknown)
Responsible Party: Principal Investigator, Marie-Rose Van Hoestenberghe, MD, Neonatologist, Ziekenhuis Oost-Limburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B331201422729
Record Dates: First submitted 2017-02-16; First posted 2017-07-27 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Premature Birth
Keywords: prematurity; psychomotor development; parent empowerment; e-health; parental support; post discharge follow-up
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- INTNIC (Experimental): NICU Intervention Group Web Application Infants < 32 weeks
  Interventions: Other: Web Application
- CNIC (No Intervention): NICU Control Group No Web Application Infants < 32 weeks
- CMAT (No Intervention): Maternity Unit Control Group No Web Application Infants > 37 weeks

INTERVENTIONS:
Other: Web Application — Parents receive a web application that offers information and support until the age of 2.
  Arms: INTNIC

SUMMARY:
The main purpose of the neonatal intensive care unit (NICU) is to optimize the development of the newborn. Preterm children are at greater risk for developmental disorders. On the one hand, this is due to cerebral complications inherent to the prematurity, on the other hand it is related to the very early and therefore vulnerable stage of brain development at the time of the premature birth. The development of the child is also the result of a constant interaction between the infant and its environment, primarily the primary caregiver (i.e. the parents). A premature birth can cause great stress to parents, and there are several obstacles that can make it difficult to handle their child. Therefore, we have developed a web application that supports parents until their child reaches the age of two. By keeping them informed, we hope to make them more confident in their role as parents, and thus facilitate the parent-child interaction. In order to determine whether this form of support has an additional effect on the development of the premature child, we compare two groups of premature infants and a group of non-premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Premature birth (< 32 weeks)

Exclusion Criteria:

* The lack of internet access or a personal email account
* Little or no knowledge of Dutch in both parents
* Children with a congenital disease

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2014-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Bayley-III-NL | 5 months, 1 year, 2 year
  Bayley Scales of Infant and Toddler Development Mental, social and motor development of the child
Change in DT-P | 2 weeks after birth, 37 weeks PMA, 5 months, 1 year, 2 year, 5 year
  Distress Thermometer for Parents
Change in EMPO | 2 weeks after birth, 37 weeks PMA, 5 months, 1 year, 2 year, 5 year
  Dutch Empowerment Questionnaire Parental empowerment in raising children (intrapersonal, interactional, and behavioral)
WPPSI-III-NL | 5 year
  Wechsler Preschool and Primary Scale of Intelligence Cognitive Development of the Child

SECONDARY OUTCOMES:
Change in PNAR | 2 weeks after birth, 37 weeks PMA, 5 months, 1 year, 2 year, 5 year
  Parent Newborn Attachment Relationship Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Rose Van Hoestenberghe, MD., Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Schiepse Bos 6, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No